CLINICAL TRIAL: NCT01047215
Title: Changes of Heart Rate Variability in Schizophrenic and Bipolar Patients Under the Medication of Aripiprazole and Quetiapine
Brief Title: Heart Rate Changes in Schizophrenic and Bipolar Patients Under the Medication of Aripiprazole and Quetiapine
Acronym: HeartAriQue
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: IRB TCVGH, Taichung Veterans General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C09032
Record Dates: First submitted 2010-01-06; First posted 2010-01-12 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Schizophrenia; Bipolar
Keywords: schizophrenia; bipolar; aripiprazole; quetiapine
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole; Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aripipazole (Active Comparator): Heart rate change in schizophrenic and bipolar patients under the aripipazole and quetiapine medication
  Interventions: Drug: Aripiprazole; Quetiapine
- Quetiapine (Active Comparator): Heart rate change in schizophrenic and bipolar patients under the aripipazole and quetiapine medication
  Interventions: Drug: Aripiprazole; Quetiapine

INTERVENTIONS:
Drug: Aripiprazole; Quetiapine — Aripiprazole Quetiapine

SUMMARY:
The goal of this research is investigating the heart rate changes in schizophrenic and bipolar patients under the medication of aripiprazole and quetiapine. In the mean time, we are hoping further investigating the interrelationship of medicine dosage and heart rate change, in order to acquire the best relationship both effectiveness as well as safety in acceptable heart rate change of clinical suggestion.

DETAILED DESCRIPTION:
Primary Goal: The goal of this research is investigating the heart rate changes in schizophrenic and bipolar patients under the medication of aripiprazole and quetiapine. As we known, clozapine, an antipsychotic, could cause fatal cardiac arrhythmia; in previous reports showed fatal rate about 0.7%, in spite of not very high, it reflects heart rate change decreasing. Therefore, many researches begin to focus on the relationship and heart rate change. Quetiapine, an atypical antipsychotic, FDA approved in 1997, Department of Health (DOH) in Taiwan also approved for schizophrenia for its effectiveness of negative disorders, low extrapyramidal syndrome, low side-effects of muscle catatonia and sluggishness. The side-effects of quetiapine are lethargy, nausea (occur rate 9%-44%), insomnia (12%), postural hypotension (4%-7%), constipation(8-10%), thirsty (9%-44%), weight gain (5-23%) and liver enzyme (GGT、AST、ALT) increasing (6%). Aripiprazole, FDA approved in 2002, DOH in Taiwan also approved for schizophrenia for its effective remittance of positive disorders, also effective for negative disorders and cognitive function regression. Besides, aripiprazole combine lithium or valproic acid can control the onset of manic and mixure of bipolar patients. The side-effects of aripiprazole are few, low extrapyramidal syndrome, no significant weight gain and blood sugar level, not surge in prolactin level and low menstrual cycle abnormal, gynecomastia and sexual dysfunction. Other side-effects are postural hypotension (0.6%-4%), headache (12%-27%), lethargy (8%-18%), insomnia (5%-26.3%), constipation (5-11%). Both quetiapine and aripiprazole are atypical antipsychotic, serious side-effects are fewer than typical antipsychotics, however, in some sensitive patients still have some side-effects such as limb-stiffness and akathisia (quetiapine 4%-12%, aripiprazole 2%-27.3%). In some retrospect researches, quetiapine will increase the opportunity of cardio- sudden death and pass off by 0.3%-1% in age 30-74 adult. On the other hand, aripiprazole (0.1%-1%) showed prolonging of QT wave which was considered as a danger factor of fatal arrhythmia. Despite of the danger, serious side-effects are rare, aripiprazole and quetiapine are widely used in clinical.

This study hope to further study whether quetiapine and aripiprazole will occur heart rate changes similar to clozapine, using heart rate changes approach to find out the possibility of causing arrhythmia and fatal of these 2 medicines.

Secondary goal:

1. Further investigate the relationship of drug dosage and heart rate change, in order to acquire the best relationship both effectiveness as well as safety in acceptable heart rate change of clinical suggestion.
2. The subjects of this study are schizophrenic and bipolar patients, who use quetiapine and aripiprazole, also will stratify into gender, age and influence of heart rate changes.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 to 50, all genders.
2. Psychiatry doctor diagnosed who met DSM-IV-TR criteria schizophrenia or bipolar patients and using antipsychotics.
3. Psychiatry doctor first diagnosed who met DSM-IV-TR criteria schizophrenia or bipolar patients and without using antipsychotics.
4. Participants understand the goal of this experiment and willing to cooperate for evaluating heart rate change measurement. Participants need to understand the procedure of this study.
5. Participants voluntarily join this interview, approximately 30-45min.
6. Clinical reviewed patient's condition need to use quetiapine or aripiprazole.

Control group

1. Age between 20 to 50, all genders.
2. Psychiatry doctor diagnosed who exclude DSM-IV-TR schizophrenia or bipolar patients.
3. Participants understand the goal of this experiment and willing to cooperate for evaluating heart rate change measurement. Participants need to understand the procedure of this study.
4. Participants voluntarily join this interview, approximately 30-45min.

Exclusion Criteria:

Experimential Group:

1. Participants fail to understand the goal of this experiment and unwilling to cooperate for evaluating heart rate change measurement.
2. Participant has another major mental disease other than the inclusion criteria.
3. Participants have cardio-vascular disease, diabetes, hepatic cirrhosis, kidney disease, material abuser (smoking not excluded) and long-term-effective psychotics user.
4. Participant has combination diseases, it could seriously influence diagnosis.
5. Psychopathy or psychosis can not be categorized in defined group.
6. Clinical reviewed patient's condition need to switch other medicine.
7. Clinical reviewed patient's condition need to quite this experiment and record reasons.
8. Participants decide to quite experiment without any conditions.

Control group

1. Participants fail to understand the goal of this experiment and unwilling to cooperate for evaluating heart rate change measurement.
2. Participants have cardio-vascular disease, diabetes, hepatic cirrhosis, kidney disease, material abuser (smoking not excluded) and long-term-effective psychotics user.
3. Participants decide to quite experiment without any conditions.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-08; Primary Completion 2009-08 (Actual); Study Completion 2010-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tsuo-Hung Lan, MD., PhD., Study Director — Taichung Veterans General Hospital; Tsuo-Hung Lan, MD.,PhD, Study Director — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan, Taiwan